## STATISTICAL ANALYSIS PLAN FOR: Soft Exosuits for Functional Gait Recovery in Acute Stroke Rehabilitation (NCT06231511) Last Updated: 5/15/2025

Statistical Methods for Primary Outcome Measure:

For each study arm, descriptive statistics were used to summarize the primary outcome measure. Specifically, the mean and range (minimum and maximum values) were calculated and reported to characterize the distribution of outcomes within each arm. No formal hypothesis testing was conducted.